CLINICAL TRIAL: NCT02279706
Title: Linguistic Adaptation of Rhinitis Control Assessment Test (RCAT) in Korean and Responsiveness to Disease Severity, Quality of Life, and Treatment in Adult Rhinitis Patients: A Multicenter Prospective Study
Brief Title: Korean Linguistic Adaptation of Rhinitis Controlled Assessment Test
Acronym: R-CAT
Status: Completed | Type: Observational
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Hae-Sim Park, professor, Department of allergic interal medicine, Ajou University School of Medicine
Other Study IDs: MED-OBS-14-158
Record Dates: First submitted 2014-10-17; First posted 2014-10-31 (Estimated); Last update posted 2016-05-02 (Estimated); Status verified 2016-04

CONDITIONS: Rhinitis
MeSH Terms: conditions — Rhinitis | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: questionnaire — Check the Korean version of rhinitis controlled assessment tests, the total non-symptom scores (total nasal symptoms score, TNSS), rhinitis-related quality of life (RQLQ), rhinitis controlled degree, severity, and after study enrollment and 4 weeks treatment.
  Other Names: questionnaire(R-CAT-RQLQ)

SUMMARY:
Korean linguistic adaptation of Rhinitis controlled assessment test (RCAT).

DETAILED DESCRIPTION:
Check the Korean version of rhinitis controlled assessment tests, the total non-symptom scores (total nasal symptoms score, TNSS), rhinitis-related quality of life (RQLQ), rhinitis controlled degree, severity, and after study enrollment and 4 weeks treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Adults over 19 years
2. Past medical history and allergy skin test or who have been diagnosed with allergic or non-allergic rhinitis, based on serum specific immunoglobulin E .
3. People who have experienced symptoms of rhinitis within 12 months from the time of study enrollment.
4. People who have rhinitis symptoms requiring medication at the time of study enrollment.
5. People who can read and write korea language.
6. People who signed a written consent form approved by the Institutional Review Board of their respective organizations to participate in this study freely hearing to explain fully the purpose for the contents of this study prior to participation in research.

Exclusion Criteria:

1. People diagnosed with Rhinitis medicamentosa.
2. People determined that bacterial or viral respiratory infection at the time of study enrollment.
3. People who have evidence of nasal infection
4. People associated anatomical abnormality that causes severe nasal congestion as deviation of nasal septum.
5. People determined that acute or chronic sinusitis according to the researchers determined.
6. In case that pregnancy test is positive, or ambiguous conclusions among female patients.
7. people deemed unsuitable for clinical trial participation due to other reasons.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: rhinitis within 12 months from the time of study enrollment.
Sampling Method: Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2014-10; Primary Completion 2015-09 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Korean linguistic adaptation of Rhinitis controlled assessment test (RCAT) | up to 4weeks
  Check the Korean version of rhinitis controlled assessment tests

SECONDARY OUTCOMES:
rhinitis-related quality of life | up to 4weeks
  rhinitis-related quality of life (RQLQ)check up to 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: hae sim park, professor, Principal Investigator — Department of internal medicine
Locations (1):
- Ajou University Medical Center, Suwon, South Korea